CLINICAL TRIAL: NCT07173270
Title: Improved Oral Health in Head and Neck Cancer Survivors
Acronym: OHHNC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Region Västerbotten (Other Government); Region Östergötland (Other); Sjöbergstiftelsen (Unknown); The Stig & Ragna Gorthon Foundation, Helsingborg (Unknown); Swedish Cancer Society (Other); Region of Uppsala (Unknown); Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-05510-01
Record Dates: First submitted 2025-08-26; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer Squamous Cell Carcinoma; Head and Neck Cancer
Keywords: Head and neck cancer; Nutrition; Oral health; cancer survivors; Quality of Life; healthcare costs
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral health intervention (Other): The intervention group will receive examination and treatment by a dental hygienist every 3 months starting 6 months after completion of RT/CRT up to 3 years.
  Interventions: Other: Oral health support

INTERVENTIONS:
Other: Oral health support — The intervention group will receive examination and treatment by a dental hygienist every 3 months starting 6 months after completion of RT/CRT up to 3 years. During visits to the dental hygienist, they will be asked about oral hygiene habits, fluoride use, dry mouth problems, and dietary habits (including intake of easily degradable carbohydrates). Oral dryness will be assessed using the Clinical Oral Dryness Scale. The stimulated salivary secretion and buffering capacity will be assessed, and the ability to open the mouth, cariological and periodontal status and registered plaque. Based on the results of the clinical examination, the patient will get individually tailored advice and recommendations on oral hygiene, fluoride use, dry mouth relief, and support in reducing the intake of food items and drinks with high sugar content. Professional oral care will be given, and fluoride applications when indicated.

SUMMARY:
The goal of this clinical trial is to learn if an oral care programme can prevent or reduce late oral side effects in patients with head and neck cancer following treatment. The main questions it aims to answer are:

* Can additional support from hospital dental care for cancer survivors, up to three years after completion of treatment, improve patients' oral health, nutritional status, quality of life, and reduce stress and anxiety compared to standard care?
* Are there differences in oral health outcomes between younger and older individuals receiving additional support from hospital dental care?
* Can additional support from hospital dental care for cancer survivors, up to three years after completion of treatment, reduce the duration of sick leave and enhance patients' ability to return to work compared to standard care?
* Can additional support from hospital dental care for cancer survivors, up to five years after completion of treatment, be cost-effective from a health economic perspective?

Researchers will compare oral care programme to standard care to see if the programme works to improve oral health, reduce oral symptoms and problems, enhance quality of life and lower the economic costs of healthcare

Participants will:

Participate in an oral care programme, every three months for three years.

DETAILED DESCRIPTION:
In Sweden, approximately 1,800 individuals are diagnosed with head and neck cancer (HNC) each year. Treatment includes radiotherapy or surgery, sometimes combined with chemotherapy. The five-year survival rate for the entire group is now approximately 70%. Despite improved five-year survival during the last two decades, side effects such as decreased salivation, difficulty swallowing, pain and radiation-induced caries are common, which negatively affect quality of life. Thus, therapeutic improvements that support oral health are highly demanded among the large group surviving head and neck cancer. The research project is a multicentre randomised controlled trial evaluating the effectiveness of an oral care programme in preventing or reducing late oral side effects in patients with HNC following treatment. Through a collaborative effort across five healthcare regions, this study aims to provide robust evidence of the efficacy of interventions designed to improve oral health outcomes and enhance the overall quality of life among head and neck cancer survivors. The intervention group will visit a dental hygienist every 3 months for oral health examination and treatment, whereas the control group will receive standard care (i.e., they will contact dental care on their own, if needed). Data collection will include patient-reported outcome measures, nutritional status, oral and dental assessments, as well as saliva and blood samples. The goal is to enhance the understanding of how oral health and quality of life can be improved in this vulnerable group, as well as how health economic costs can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* patients (≥ 18 years)
* diagnosed with HNC
* scheduled for treatment with curative intent, including RT or CRT with or without surgery

Exclusion Criteria:

* severe alcoholism
* cognitive impairment
* inability to understand the Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-24 (Estimated); Primary Completion 2035-05-31 (Estimated); Study Completion 2045-09-23 (Estimated)

PRIMARY OUTCOMES:
Number of remaining teeth | Data will be collected before RT/CRT begins (baseline), at 6 months after the completion of RT/CRT (randomisation, start of intervention), and at one, two and three years
Maximum interincisal opening (MIO) | Data will be collected before RT/CRT begins (baseline), at 6 months after the completion of RT/CRT (randomisation, start of intervention), and at one, two and three years
Presence of caries | Data will be collected before RT/CRT begins (baseline), at 6 months after the completion of RT/CRT (randomisation, start of intervention), and at one, two and three years
Loss of supporting tissue (periodontitis) | Data will be collected before RT/CRT begins (baseline), at 6 months after the completion of RT/CRT (randomisation, start of intervention), and at one, two and three years
Osteoradionecrosis. | Data will be collected before RT/CRT begins (baseline), at 6 months after the completion of RT/CRT (randomisation, start of intervention), and at one, two and three years

SECONDARY OUTCOMES:
Health-related quality of life | Data will be collected before RT/CRT begins (baseline), at 6 months after the completion of RT/CRT (randomisation, start of intervention), and at one, two and three years.
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30. Developed by the European Organization for Research and Treatment of Cancer. General questionnaire for patients with cancer, 30 questions. Measures physical, role, emotional, cognitive and social functioning. One question about overall quality of life and nine questions about various symptoms, such as fatigue, pain and sleep difficulties. Likert scale with four response options. A higher score suggests a better level of functioning, while a higher score suggests more severe problems regarding symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No